CLINICAL TRIAL: NCT01156038
Title: Atopy Patch Test in Normal Population : Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Mahidol University, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 599/2552(EC4)
Record Dates: First submitted 2010-05-16; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Normal
Keywords: Atopy patch test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atopy patch test (Experimental): Atopy patches were applied on healthy volunteer's back for 48 hrs then the patches were removed. Reaction was evaluated 48 and 72 hrs after applying atopy patch test
  Interventions: Device: Atopy patch test with food allergen

INTERVENTIONS:
Device: Atopy patch test with food allergen — Atopy patches used with food lyophilized allergen and commercial allergen were placed on back of subjects for 48 hrs then atopy patches were taken off. Subjects should return to evaluate reaction one day later(72 hrs after applying atopy patch test)

SUMMARY:
Atopy patch test in normal population

DETAILED DESCRIPTION:
The initial diagnostic work up of suspected food allergy includes patient's history, skin prick test (SPT), measurement of food specific immunoglobulin E (IgE) with serological assays, and more recently the atopy patch test. A positive SPT seems to reflect early reactions to food challenges, whereas the atopy patch test has a high diagnostic efficacy for late phase clinical reactions. The purpose of this study was to evaluate atopy patch test reaction in non-atopic population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age 18-40 yrs
* Volunteer sign for informed consent

Exclusion Criteria:

* who have dermographism
* who have chronic disease eg.autoimmune disease, immune deficiency, cancer or allergic disease
* pregnant women
* who have severe eczema
* who receive antihistamine, topical steroid and systemic steroid > 20 mg/day within 7 days prior study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Reaction of atopy patch test | 3 days
  To evaluate outcome of atopy patch test reaction in non-atopic subject

SECONDARY OUTCOMES:
Comparisons atopy patch test reaction between lyophilized allergen and commercial allergen | 3 days
  To compare outcome of atopy patch test reaction using lyophilized allergen and commercial allergen

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, Professor, Study Director — Mahidol University
Locations (1):
- Department of Pediatrics, Siriraj hospital, Mahidol University, Bangkok, Thailand